CLINICAL TRIAL: NCT00354783
Title: Continuity of Leg Movements in VLBW Premature Infants: From Spontaneous Kicking and Supported Stepping to Independent Walking
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361701209
Record Dates: First submitted 2006-07-18; First posted 2006-07-20 (Estimated); Last update posted 2006-07-20 (Estimated); Status verified 2006-07

CONDITIONS: Premature Birth
Keywords: Very low birth weight premature infants; Kicking; Stepping; Walking; Motor development; Kinematics
MeSH Terms: conditions — Premature Birth; Gait Disorders, Neurologic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
The purposes of this one-year follow-up study are twofold: (1) to prospectively examine the spontaneous kicking and the supported stepping movement in VLBW premature infants until attainment of independent walking; and (2) to assess factors (i.e. gross motor development, cardiopulmonary function, anthropometry, body composition and cognition) that could potentially influence walking attainment in VLBW premature infants.

DETAILED DESCRIPTION:
Very low birth weight (VLBW) preterm infants (birth weight < 1,500g) sustain a high risk of neuromotor disability, as exemplified by delayed walking attainment. Spontaneous kicking and supported stepping have been proposed as the early precursors to independent walking. The continuity of these early leg movements with independent walking has been established in normal term infants, but such relations remain unclear in VLBE premature infants. Therefore, the purposes of this one-year follow-up study are twofold: (1) to prospectively examine the spontaneous kicking and the supported stepping movement in VLBW premature infants until attainment of independent walking; and (2) to assess factors (i.e. gross motor development, cardiopulmonary function, anthropometry, body composition and cognition) that could potentially influence walking attainment in VLBW premature infants. This study will enroll 15 VLBW premature infants born at National Taiwan University Hospital. Infants will be scheduled for spontaneous kicking examination at 2 and 4 months of corrected age, followed by supported stepping examination at 9 and 11 months of corrected age and recorded their age of walking attainment. Age of walking attainment is defined as the time when the child is first able to move for five successive steps without support. At each visit, infants will be examined for spontaneous kicking or supported stepping movements (with three-dimensional kinematic analysis of Peak Motion Analysis System), gross motor function (with the Alberta Infant Motor Scale), cardiopulmonary function (with a pulsed oxymeter), anthropometry (with scale and tape measure), body composition (with the Pediatric Plicometric System) and cognition (with the Chinese Child Development Inventory- Cognitive Subscale). The results of this study will provide important information to help reveal the maturation process of early leg movements prior to walking attainment in premature infants. Furthermore, the identified early neuromotor markers and influencing factors for walking attainment will provide physical therapists useful guidance in making early treatment plans for those premature infants who will develop motor delays.

ELIGIBILITY:
Inclusion Criteria:

* BW below 1500 gm
* GA under 37 weeks

Exclusion Criteria:

* Existence of congenital anomalies and genetic disease

Ages: 0 Years to 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15
Dates: Start 2007-01; Study Completion 2007-12

CONTACTS AND LOCATIONS:
Overall Officials: Suh-Fang Jeng, Sc.D, Study Director — National Taiwan University